CLINICAL TRIAL: NCT06929338
Title: A Feasibility Study to Evaluate a Precision Oncology Platform (xDRIVE) in Participants With Advanced Colorectal Cancer
Brief Title: xDRIVE in Metastatic Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: First Ascent Biomedical Inc. (Industry)
Collaborators: Mayo Clinic (Other); Florida International University (Other)
Responsible Party: Sponsor
Other Study IDs: FAB00000001
Record Dates: First submitted 2025-03-27; First posted 2025-04-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Colon Cancer; Metastatic Rectal Adenocarcinoma; Metastatic Rectal Carcinoma; Metastatic Rectum Cancer
Keywords: functional precision medicine; artificial intelligence; molecular tumor profiling; metastatic colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Live tumor tissue samples with DNA and RNA isolated for tumor profiling and treatment identification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic colorectal cancer patients: Participants with mCRC who need clinical tumor biopsy or resection and need to start systemic therapy for measurable disease.
  Interventions: Diagnostic Test: Functional precision medicine

INTERVENTIONS:
Diagnostic Test: Functional precision medicine — The results of the drug sensitivity assay and genetic screening will be used to inform treating physician about patient-specific drug sensitivity or resistance guiding best therapy choices. Treatment will not be given as part of the study.

SUMMARY:
The study aims to evaluate the clinical utility of the xDRIVE functional precision medicine + artificial intelligence (AI) platform in predicting treatment response for metastatic colorectal cancer (mCRC). The primary objective is to assess xDRIVE's accuracy in forecasting clinical benefit from standard-of-care (SOC) therapies, with a target of ≥80% accuracy in 25 participants. Achieving this threshold would provide sufficient statistical power to reject the null hypothesis of ≤50% accuracy.

The secondary goal is to determine the feasibility of utilizing xDRIVE for timely treatment recommendations. Success will be defined by the ability to provide recommendations within four weeks for at least 64% of patients, ensuring clinical applicability.

Additionally, the study includes an exploratory objective to examine oncologists' perspectives on integrating xDRIVE into clinical decision-making. This will be achieved through a post-hoc survey assessing physician experiences with the precision oncology platform.

DETAILED DESCRIPTION:
Metastatic colorectal cancer (mCRC) remains a critical unmet clinical need, necessitating innovative approaches to improve patient outcomes. Functional precision medicine (FPM)-guided interventions offer the potential to enhance treatment decision-making by tailoring therapies based on individual patient responses. This study aims to evaluate the clinical utility of xDRIVE, a precision oncology platform, in predicting treatment response to standard-of-care (SOC) therapies in patients with advanced colorectal cancer. By integrating cutting-edge biobanking and personalized medicine approaches, the study seeks to determine whether xDRIVE can provide accurate and timely treatment recommendations, ultimately optimizing clinical management for patients with mCRC.

The primary objective is to assess the accuracy of xDRIVE in predicting clinical benefit, defined as a complete response, partial response, or stable disease. Success will be determined by achieving at least 80% accuracy in 20 of 25 participants, allowing for rejection of the null hypothesis (≤50% accuracy) with 90% statistical power. A total of 30 participants will be enrolled to ensure robust evaluation. The secondary objective is to evaluate the feasibility of utilizing xDRIVE in a clinically actionable timeframe, with success defined as delivering treatment recommendations within four weeks for at least 64% of cases. This feasibility threshold will allow for rejection of the null hypothesis (≤35% feasibility) with 90% power. Additionally, the study will explore oncologists' perspectives on integrating xDRIVE into clinical decision-making. A post-hoc survey will be conducted to assess physician experiences, providing insights into the potential impact and adoption of precision oncology platforms in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants (men and women) enrolled in internal review board (IRB) 622-00 and meet the following criteria.
* Participants ≥18 years of age with a diagnosis of mCRC who are willing to consent to the study
* Participants with Eastern Cooperative Group (ECOG) performance status of 0, 1, or 2.
* Participants with measurable disease
* Participants who need to start SOC cancer-directed systemic therapy
* Participants able to provide treatment and outcome information from previous lines of therapy.
* Participants who will need a tumor biopsy, excision, or resection as part of their routine clinical care.
* Participants willing to have a blood draw performed for matched normal material.
* Participants who plan to have their first radiographic assessment of their cancer at Mayo Clinic.

Exclusion Criteria:

* Participants who do not have malignant tissue available or safely accessible or do not have sufficient amount of tissue from anticipated biopsy, excision or resection for testing.
* Participants who do not have measurable disease.
* Participants with insufficient health indicators to undergo therapeutic intervention for mCRC based on treating oncologist's clinical assessment.
* Participants with other concurrent cancers besides mCRC which also require ongoing cancer-directed therapy.
* Participants who cannot provide an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with mCRC who need clinical tumor biopsy or resection and need to start systemic therapy for measurable disease.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Accurate prediction of clinical benefit (complete response, partial response or stable disease) to physician-selected treatment among among enrolled patients with mCRC | Tumor measurements will be taken at baseline before treatment and at the first post-treatment scan. RECIST will be used to assess response. Outcomes will be tracked for the duration of the study, up to one year.
  The primary objective is to determine the accuracy of clinical benefit prediction by xDRIVE testing in participants with advanced CRC who receive SOC therapies. Response to SOC therapy will be determined by RECIST guidelines, with disease response measured through radiographic imaging.
  Accurate prediction of RECIST-determined clinical response (complete response, partial response, stable disease, or progressive disease) by xDRIVE tumor in 20 of 25 participants (80%) is sufficient to reject the null hypothesis (≤50% accuracy) with 90% power (α = 0.05).
  Enrollment will be a total of 30 subjects.

SECONDARY OUTCOMES:
Feasibility of returning xDRIVE functional precision medicine data in a clinically-actionable timeframe | Timeframe for successful return of data is within 4 weeks. Previous studies have demonstrated a median 10-day turnaround time.
  The secondary objective is to determine the feasibility of using xDRIVE to provide treatment recommendation in a clinically-actionable timeframe. Feasibility will be demonstrated if treatment recommendations are returned within 4 weeks for at least 16 of 25 patients (64%), which is sufficient to reject the null hypothesis (≤35% treatment recommendations) with 90% power (α = 0.05).

OTHER OUTCOMES:
Assessment of physician experience with xDRIVE functional precision medicine through post-hoc questionnaire | Post-hoc questionnaire will initiated at baseline and will be completed within 2 weeks following radiographic imaging of patient response. Questionnaires will be performed on a per-participating physician basis.
  The exploratory objective is to assess treating oncologists' perspective on the use of precision oncology platform in participants with advanced CRC, investigated through a post-hoc questionnaire of physician experience.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Berlow, PhD, Principal Investigator — First Ascent Biomedical; Hao Xie, MD PhD, Principal Investigator — Mayo Clinic; Lisa Boardman, MD, Principal Investigator — Mayo Clinic; Diana J Azzam, PhD, Principal Investigator — Florida International University

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will be kept only at the clinical site and only for the purpose of tracking patient enrollment and outcomes, and will not be shared even with other sites in the study.

REFERENCES:
- [Background] Acanda de la Rocha AM, Berlow NE, Azzam DJ. Functional precision medicine: the future of cancer care. Trends Mol Med. 2025 May;31(5):404-408. doi: 10.1016/j.molmed.2024.10.015. Epub 2024 Nov 19. PMID 39567286
- [Background] Acanda De La Rocha AM, Berlow NE, Fader M, Coats ER, Saghira C, Espinal PS, Galano J, Khatib Z, Abdella H, Maher OM, Vorontsova Y, Andrade-Feraud CM, Daccache A, Jacome A, Reis V, Holcomb B, Ghurani Y, Rimblas L, Guilarte TR, Hu N, Salyakina D, Azzam DJ. Feasibility of functional precision medicine for guiding treatment of relapsed or refractory pediatric cancers. Nat Med. 2024 Apr;30(4):990-1000. doi: 10.1038/s41591-024-02848-4. Epub 2024 Apr 11. PMID 38605166